CLINICAL TRIAL: NCT00841438
Title: Efficacy of Clotinab in Acute Myocardial Infarction Trial- ST Elevation Myocardial Infarction
Brief Title: Efficacy of Early Administration of Clotinab in Acute Myocardial Infarction
Acronym: ECLAT-STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: ISU ABXIS (Korea pharmaceutical company) (Unknown)
Responsible Party: Yangsoo Jang, Severance hospital, Yonsei university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISU-CLT-07001
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-02

CONDITIONS: Myocardial Infarction
Keywords: Angioplasty; Transluminal; Percutaneous Coronary
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Provisional use of Clotinab (Active Comparator): Provisional use of clotinab
  Interventions: Drug: Clotinab
- Upstream use of clotinab (Experimental): early upstream use of clotinab
  Interventions: Drug: Clotinab

INTERVENTIONS:
Drug: Clotinab — Clotinab: IV bolus 0.25 mg per Kg and a 12-hour IV infusion 0.125 μg per kg
  Other Names: Clotinab, Gp IIb/IIIa inhibitor
  Arms: Provisional use of Clotinab
Drug: Clotinab — Clotinab: IV bolus 0.25 mg per Kg and a 12-hour IV infusion 0.125 μg per kg
  Other Names: Clotinab, Gp IIb/IIIa inhibitor
  Arms: Upstream use of clotinab

SUMMARY:
The ADMIRAL (Platelet glycoprotein IIb/IIIa inhibition with coronary stenting for acute myocardial infarction) study demonstrated that early administration of abciximab in patients with ST elevation acute myocardial infarction prior to PCI improves clinical outcomes but no specifically designed randomized study has addressed the issue of early upstream use of GP IIb/IIIa inhibitors in ST elevation acute myocardial infarction who are undergoing PCI, especially in the era of routine pretreatment with 600 mg of clopidogrel. Therefore, the objective of the randomized ECLAT-STEMI study was to assess the hypothesis that the early upstream use of Clotinab is a useful therapy in patients with ST elevation MI undergoing PCI compared to "provisional use", even after pretreatment with a 600-mg loading dose of clopidogrel.

DETAILED DESCRIPTION:
It is well known that platelet-mediated thrombosis is account for the pathophysiology of acute coronary syndrome (ACS) (1,2). In the treatment of ACS, intravenous platelet glycoprotein (GP) IIb/IIIa receptor antagonists for platelet aggregation may reduce the risk of ischemic complications (3-7). Therefore, in the management of ACS, Platelet GP IIb/IIIa receptor inhibitors have been developed as a promising new therapy for the reduction of coronary events and the improvement of clinical outcomes.

Abciximab, one of platelet GP IIb/IIIa receptor blockers, was developed by Coller in 1985 and named as 7E3(8). Abciximab is a chimeric human monoclonal antibody and binds to platelet surface GP IIb/IIIa receptor competitively with adhesive molecules such as fibrinogen and von Willebrand factor, and blocks the final stage of platelet aggregation(9). The effect of Abciximab has been proved in many clinical trials such as the EPIC trial(9), EPILOG trial(10), TARGET(11) etc. The contribution of GP IIb/IIIa inhibition in ACS (Tirofiban) is shown in placebo-controlled trials in which upstream GP IIb/IIIa inhibition was initiated upon admission (12,13). Although these results are encouraging, there are few other data to support the use of upstream GP IIb/IIIa inhibitors. Moreover, according to the GUSTO-IV trial (14), the use of Abciximab was not recommended in the manner of upstream use. To evaluate the role of abciximab in conservatively treated non-ST-elevation ACS patients, the GUSTO-IV study randomized 7800 patients with non-ST-elevation ACS to receive either placebo or an Abciximab bolus (0.25 mg/kg) and 24-hour or 48-hour infusion(0.125 µg/kg/min). However, in fact, a trend was noted for potential harm with the higher abciximab dose. Even subgroup analyses including high-risk troponin-positive patients showed no benefit with either abciximab regimen (9.7% with placebo, 10.2% with 24-hour abciximab, 11.7% with 48-hour abciximab for death or MI at 30 days, P = NS). Because of these results, the majority of patients received abciximab relatively late, at the time of PCI in clinical practices.

However, the ADMIRAL study (3) demonstrated that early administration of abciximab in patients with ST elevation acute myocardial infarction prior to PCI improves clinical outcomes and also no specifically designed randomized study has addressed the issue of early upstream use of GP IIb/IIIa inhibitors in ST elevation acute myocardial infarction who are undergoing PCI, especially in the era of routine pretreatment with 600 mg of clopidogrel. Therefore, the objective of the randomized ECLAT-STEMI study was to assess the hypothesis that the early upstream use of Clotinab is a useful therapy in patients with ST elevation MI undergoing PCI compared to "provisional use", even after pretreatment with a 600-mg loading dose of clopidogrel.

The Clotinab, a product made in ISU ABXIS CO., LTD, was produced by inserting anti- platelet GP IIb/IIIa DNA into Chinese hamster's ovary cell. Since it contains identical active ingredient as ReoPro® on the domestic market, it is expected that the Clotinab has same efficacy to ReoPro® as a platelet GP IIb/IIIa receptor inhibitor. Recently, the Clotinab is shown to be safe and effective in preventing ischemic heart complications for high-risk patients who will undergo PCI.

2. Study Protocol 2-1. Objectives: Randomized, controlled, single blind, multi-center trial To assess the hypothesis that the early upstream use of Clotinab is a useful therapy in patients with ST elevation myocardial infarction undergoing PCI compared to "provisional use", even after pretreatment with a 600-mg loading dose of clopidogrel.

2-2. Study Design: Efficacy of CLotinab in ST-elevation Acute myocardial infarction Trial - ST Elevation Myocardial Infarction (The ECLAT - STEMI study)

2-3. Study Endpoints:

1. Primary Endpoint: Efficacy To evaluate the effect of early upstream use of Clotinab (started at emergency room) co-administered with clopidogrel loading dose 600mg in STEMI

   - 30 Days MACCE (death, MI, TVR, cerebrovascular event)
2. Secondary Endpoint: Efficacy and Safety To evaluate the safety of early upstream use of Clotinab (started at emergency room) co-administered with clopidogrel loading dose 600mg in STEMI

   * TIMI flow at before and after PCI
   * Corrected TIMI frame count after PCI
   * Procedural success (No reflow incidence)
   * MACCE at 9 month
   * Major bleeding event (According to TIMI criteria)
   * 9 month Angiography Finding

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18-80 years of age.
2. The patient had the symptoms of acute myocardial infarction within 12 hours with ST segment elevation of more than 1 mm in at least two contiguous leads of EKG or new onset LBBB.
3. The patient or guardian agrees to the study protocol and provides informed, written consent.

Exclusion Criteria:

1. Patients to whom PCI can not be undergone within 12 hours from receiving the study drug
2. Cardiogenic shock or symptomatic hypotension or sitting SBP < 95 mmHg
3. The history of major surgery, trauma, retinal hemorrhage, significant gastrointestinal or genitourinary bleeding within recent 6 weeks;
4. History of cerebrovascular attack within two years, or cerebrovascular attack with a significant residual neurological deficit
5. Severe or malignant hypertension (= sitting SBP > 180 mmHg and/or sitting DBP > 105 mmHg)
6. The patients who require oral anticoagulants during the trial; patients who have been administrated oral anticoagulants within 7 days
7. The history or diagnosis of vasculitis; renal insufficiency (the level of serum creatinine is two times higher than the upper limit of normal of each center)
8. The patients who could not take anti-platelet drugs
9. The patients who might die of other disease than cardiac disease during the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
MACCE (death, MI, TVR, cerebrovascular event) | 30 days

SECONDARY OUTCOMES:
MACCE (death, MI, TVR, cerebrovascular event) | 9 months
TIMI flow at before and after PCI | Immediate post procedure
Corrected TIMI frame count after PCI | Immediate postprocedure

CONTACTS AND LOCATIONS:
Overall Officials: Yangsoo Jang, MD, Ph D, Principal Investigator — Division of Cardiology, Cardiovascular Hospital, Yonsei University
Locations (31):
- South Korea (31):
  - Dankook University Hospital, Cheonan
  - Chonbuk National University Hospital, Cheonju
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Health Insurance Corporation Ilsan Hospital, Goyang
  - Dongguk University International Hospital, Goyang
  - Myongji Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Pusan National University Hospital, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Hallym University sacred Heart Hospital, Pyungchon
  - Seoul National University Bundang Hospital, Seongnam
  - Yonsei University, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Kyung Hee University East-West Nea Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Youngdong Severance Hospital, Seoul
  - Catholic University of Korea, kangnam St. Mary's Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Eulji General Hospital, Seoul
  - Catholic University of Korea, St. Mary's Hospital, Seoul
  - Hallym University kangnam sacred Heart Hospital, Seoul
  - Gachon University Gil Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Kim JS, Park SM, Kim BK, Ko YG, Choi D, Hong MK, Seong IW, Kim BO, Gwon HC, Hong BK, Tahk SJ, Park SW, Kim CJ, Jeong MH, Yoon J, Jang Y; ECLAT-STEMI Trial investigators. Efficacy of clotinab in acute myocardial infarction trial-ST elevation myocardial infarction (ECLAT-STEMI). Circ J. 2012;76(2):405-13. doi: 10.1253/circj.cj-11-0676. Epub 2011 Dec 7. PMID 22146757